CLINICAL TRIAL: NCT01694667
Title: Effectiveness of Omega-3 Fatty Acids for the Reduction of Hyperactivity in Children With Autism Spectrum Disorder
Brief Title: Omega-3 Fatty Acids for Hyperactivity Treatment in Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00068694
Record Dates: First submitted 2012-03-26; First posted 2012-09-27 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Autism Spectrum Disorders; Hyperactivity
MeSH Terms: conditions — Autism Spectrum Disorder; Spasm | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 Fatty Acids (Active Comparator): Omega-3 Fatty Acids: Omega-3 fatty acids will be delivered in orange-flavored pudding packets (Coromega®, Vista, CA). Each packet contains 650 mg of omega-3 fatty acids, 350mg of eicosapentanoic acid (EPA), 230mg of docosahexanoic acid (DHA) and 2,000 mg of fish oil 18/12, and will be given twice daily for a daily dose of 1.3 grams of omega-3 fatty acids (and 1.1 grams of DHA + EPA
  Interventions: Drug: Omega-3 Fatty Acids
- Placebo (Placebo Comparator): Placebo packets will have same orange-flavored pudding with an identical appearance and taste, but will include safflower oil instead of the fish oil. One placebo packet will be given twice daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Omega-3 Fatty Acids — Omega-3 fatty acids will be delivered in orange-flavored pudding packets (Coromega®, Vista, CA). Each packet contains 650 mg of omega-3 fatty acids, 350mg of eicosapentanoic acid (EPA), 230mg of docosahexanoic acid (DHA) and 2,000 mg of fish oil 18/12, and will be given twice daily for a daily dose of 1.3 grams of omega-3 fatty acids (and 1.1 grams of DHA + EPA).
  Other Names: Omega-3; N-3 Fatty Acid
  Arms: Omega-3 Fatty Acids
Other: Placebo — Placebo packets will have same orange-flavored pudding as active Omega-3 fatty acids comparator with an identical appearance and taste, but will include safflower oil instead of the fish oil. One placebo packet will be given twice daily.
  Arms: Placebo

SUMMARY:
The proposed study is an internet-based, randomized, double-blind, placebo-controlled trial which will assess changes in hyperactivity in children ages five through eight with an autism spectrum disorders (ASD) and elevated levels of hyperactivity. In order to answer this question, this study will assess changes in hyperactivity as measured by the Aberrant Behavior Checklist (ABC) in children with ASD and elevated baseline levels of hyperactivity who are randomly assigned to use 1.3 grams of omega-3 fatty acids daily compared to placebo. The overwhelming majority of study procedures, including recruitment, informed consent, assessment of inclusion and exclusion criteria, and collection of baseline and outcome measures will take place over the internet.

DETAILED DESCRIPTION:
Families and caregivers of children enrolled in the IAN Research between the age 5-8 and with an established diagnosis of autism will be invited to participate in the study by e-mail. All of these families have previously given consent to be contacted about research opportunities. Families who respond to the e-mail recruitment letter will undergo a brief screening process to determine if the child has any exclusion criteria and to ensure the child is age 5-8, has an autism spectrum disorder, and has elevated baseline levels of hyperactivity. Families will undergo an on-line informed consent process including assent of the child. All participants will be given an opportunity to speak with a study team member should they have any questions about the study or the informed consent process. Participants will sign the informed consent using an electronic signature, a process that has been used previously in the IAN network and approved by the John's Hopkins Institutional Review Board (IRB). Families meeting all eligibility criteria will be randomly assigned and mailed the study medication (omega-3 or placebo) which will be administered to children by the parents twice daily for six weeks. Both the study medication and the matching placebo are an orange-flavored pudding that is specifically designed to be palatable for young children. Assessment of child hyperactivity, social functioning, and overall disease severity will be measured at baseline, three and six weeks by the parents, who will complete on-line standard questionnaires; ABC, Social Responsiveness Scale (SRS), clinical Global Impressions Scale (CGI).

Side effects will be assessed every week by e-mail, and any report of a side effect will immediately be followed-up with telephone contact from the PI. Although omega-3 fatty acids are extremely safe in the prescribed doses, the PI or another study physician will still be on call 24-hours-a-day, 7-days-a-week to speak to participants about possible adverse events or new medical problems (all enrolled families are provided with this 24-hour emergency phone contact information).

As part of the weekly e-mail reminder, parents will also be asked to log the medication that was provided to their children each day of the previous week to measure medication adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Children who are participating in Interactive Autism Network (IAN) Research Families
2. Diagnosis of (Autism Spectrum Disorders (ASD) by a professional and Social Communication Question (SCQ) score>12
3. Age 5-8
4. Aberrant Behavior Checklist - Hyperactivity subscale (ABC-H)>20

Exclusion Criteria:

1. Children in foster care and each parent must affirm that they are the biological or adoptive parent of the child
2. Allergy to fish
3. Bleeding disorder, current use of anticoagulant or anti-platelet therapy, or recent or planned surgery
4. Any major medical illness that interferes with regular school attendance
5. Current or recent (past six months) use of omega-3 fatty acid
6. Siblings with ASD

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Law, M.D., Principal Investigator — Kennedy Krieger Institute and Johns Hopkins University
Locations (1):
- This study is open to continental USA, Multiple Locations, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bent S, Hendren RL, Zandi T, Law K, Choi JE, Widjaja F, Kalb L, Nestle J, Law P. Internet-based, randomized, controlled trial of omega-3 fatty acids for hyperactivity in autism. J Am Acad Child Adolesc Psychiatry. 2014 Jun;53(6):658-66. doi: 10.1016/j.jaac.2014.01.018. Epub 2014 Mar 12. PMID 24839884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was limited to children between the ages of 5 and 8 with ASD and some verbal ability. E-mail invitations were sent to the 863 registered IAN members who met the above criteria and had given prior consent to be contacted about research opportunities between September 18, 2012 and October 31, 2012.
Pre-assignment Details: During the six-week recruitment period, 118 families expressed interest and completed the on-line screening form. Fifty-seven children from 28 states were deemed eligible and randomly assigned to study treatment.
Groups:
- Omega-3 Fatty Acids: Omega-3 fatty acids will be delivered in orange-flavored pudding packets and will be given twice daily for a daily dose of 1.3 grams of omega-3 fatty acids (and 1.1 grams of DHA + EPA).
  Omega-3 Fatty Acids: Omega-3 fatty acids will be delivered in orange-flavored pudding packets (Coromega®, Vista, CA). Each packet contains 650 mg of omega-3 fatty acids, 350mg of eicosapentanoic acid (EPA), 230mg of docosahexanoic acid (DHA) and 2,000 mg of fish oil 18/12, and will be given twice daily for a daily dose of 1.3 grams of omega-3 fatty acids (and 1.1 grams of DHA + EPA).
  29 participants allocated to this group.
- Placebo: Placebo packets will have same orange-flavored pudding with an identical appearance and taste, but will include safflower oil instead of the fish oil.
  Omega-3 Fatty Acids: Omega-3 fatty acids will be delivered in orange-flavored pudding packets (Coromega®, Vista, CA). Each packet contains 650 mg of omega-3 fatty acids, 350mg of eicosapentanoic acid (EPA), 230mg of docosahexanoic acid (DHA) and 2,000 mg of fish oil 18/12, and will be given twice daily for a daily dose of 1.3 grams of omega-3 fatty acids (and 1.1 grams of DHA + EPA).
  28 participants allocated to this group.
Period: Overall Study
Arm/Group | Omega-3 Fatty Acids | Placebo
Started | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Omega-3: Participants randomized to omega-3
- Placebo: Participants randomized to placebo
- Total: Total of all reporting groups
Arm/Group | Omega-3 | Placebo | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: months] | 88.2 (12.3) | 85.0 (13.2) | 86.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 26 | 24 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 24 | 23 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
ABC-Hyperactivity [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist - measures problem behaviors independently and commonly used in children with autism 5 subscales are included and for each higher scores are worse. Each item uses a 0 to 3 Likert scale
  Hyperactivity - 16 items, score ranges from 0-48
  Irritability - 15 items, score ranges from 0-45
  Stereotypy - 7 questions, score ranges from 0-21
  Lethargy - 16 questions, score ranges from 0-48
  Inappropriate speech - 4 questions, score ranges from 0-12
  Subscales were not combined to compute a total score.
  units on a scale | 28.4 (8.4) | 28.1 (7.6) | 28.2 (8.0)
ABC-Irritability [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist - measures problem behaviors independently and commonly used in children with autism 5 subscales are included and for each higher scores are worse. Each item uses a 0 to 3 Likert scale
  Hyperactivity - 16 items, score ranges from 0-48
  Irritability - 15 items, score ranges from 0-45
  Stereotypy - 7 questions, score ranges from 0-21
  Lethargy - 16 questions, score ranges from 0-48
  Inappropriate speech - 4 questions, score ranges from 0-12
  Subscales were not combined to compute a total score.
  units on a scale | 20.0 (8.9) | 16.8 (8.3) | 18.4 (8.7)
ABC-Stereotypy [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist - measures problem behaviors independently and commonly used in children with autism 5 subscales are included and for each higher scores are worse. Each item uses a 0 to 3 Likert scale
  Hyperactivity - 16 items, score ranges from 0-48
  Irritability - 15 items, score ranges from 0-45
  Stereotypy - 7 questions, score ranges from 0-21
  Lethargy - 16 questions, score ranges from 0-48
  Inappropriate speech - 4 questions, score ranges from 0-12
  Subscales were not combined to compute a total score.
  units on a scale | 8.0 (6.0) | 5.4 (4.7) | 6.7 (5.5)
ABC-Lethargy [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist - measures problem behaviors independently and commonly used in children with autism 5 subscales are included and for each higher scores are worse. Each item uses a 0 to 3 Likert scale
  Hyperactivity - 16 items, score ranges from 0-48
  Irritability - 15 items, score ranges from 0-45
  Stereotypy - 7 questions, score ranges from 0-21
  Lethargy - 16 questions, score ranges from 0-48
  Inappropriate speech - 4 questions, score ranges from 0-12
  Subscales were not combined to compute a total score.
  units on a scale | 12.2 (8.8) | 8.8 (4.2) | 10.5 (7.1)
ABC-Inappropriate Speech [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist - measures problem behaviors independently and commonly used in children with autism 5 subscales are included and for each higher scores are worse. Each item uses a 0 to 3 Likert scale
  Hyperactivity - 16 items, score ranges from 0-48
  Irritability - 15 items, score ranges from 0-45
  Stereotypy - 7 questions, score ranges from 0-21
  Lethargy - 16 questions, score ranges from 0-48
  Inappropriate speech - 4 questions, score ranges from 0-12
  Subscales were not combined to compute a total score.
  units on a scale | 7.0 (3.4) | 5.8 (2.8) | 6.4 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Aberrant Behavior Checklist - Hyperactivity Subscale (ABC-H) Score
Description: The Aberrant Behavior Checklist (ABC) is a 58-item survey. Items are rated on a 4-point scale from "0=no problem" to "3=major problem." Higher scores indicate greater severity. Scores can be computed for five subscales: hyperactivity, lethargy, stereotypical behavior, irritability, and inappropriate speech. The hyperactivity subscale is comprised of 16 items. The outcome measure is the change from baseline to 6 weeks. The total score ranges from 0 to 48.
Time Frame: Baseline, 6 weeks (3 week value to be collected)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 29 | 28
units on a scale | -5.3 (7.2) | -3.4 (7.5)

2. Secondary Outcome: Change in Aberrant Behavior Checklist - Lethargy Subscale Score
Description: The Aberrant Behavior Checklist (ABC) is a 58-item survey. Items are rated on a 4-point scale from "0=no problem" to "3=major problem." Higher scores indicate greater severity. Scores can be computed for five subscales: hyperactivity, lethargy, stereotypical behavior, irritability, and inappropriate speech. The lethargy subscale is comprised of 16 items. The outcome measure is the change from baseline to six weeks in the scale. Total score ranges from 0 to 48.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 29 | 28
units on a scale | -2.1 (4.2) | 0.1 (2.6)

3. Secondary Outcome: Change in Aberrant Behavior Checklist - Stereotypy Subscale Score
Description: The Aberrant Behavior Checklist (ABC) is a 58-item survey. Items are rated on a 4-point scale from "0=no problem" to "3=major problem." Higher scores indicate greater severity. Scores can be computed for five subscales: hyperactivity, lethargy, stereotypical behavior, irritability, and inappropriate speech. The stereotypy subscale is comprised of 7 items. The outcome measure is the change from baseline to six weeks in the scale. Total score ranges from 0 to 21.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 29 | 28
units on a scale | -2.0 (3.7) | -0.5 (2.6)

4. Secondary Outcome: Aberrant Behavior Checklist - Irritability Subscale Score
Description: The Aberrant Behavior Checklist (ABC) is a 58-item survey. Items are rated on a 4-point scale from "0=no problem" to "3=major problem." Higher scores indicate greater severity. Scores can be computed for five subscales: hyperactivity, lethargy, stereotypical behavior, irritability, and inappropriate speech. The irritability subscale is comprised of 15 items. The outcome measure is the change from baseline to six weeks in the scale. Total score ranges from 0 to 45.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 29 | 28
units on a scale | -2.0 (6.9) | -2.1 (4.4)

5. Secondary Outcome: Aberrant Behavior Checklist - Inappropriate Speech Subscale Score
Description: The Aberrant Behavior Checklist (ABC) is a 58-item survey. Items are rated on a 4-point scale from "0=no problem" to "3=major problem." Higher scores indicate greater severity. Scores can be computed for five subscales: hyperactivity, lethargy, stereotypical behavior, irritability, and inappropriate speech. The inappropriate speech subscale is comprised of 4 items. The outcome measure is the change from baseline to six weeks in the scale. Total score ranges from 0 to 12.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 29 | 28
units on a scale | -0.6 (2.7) | -0.9 (2.2)

6. Secondary Outcome: Change in Social Responsiveness Scale (SRS) Score
Description: Social interaction will be assessed with the SRS. This scale examines the presence and extent of autistic social impairment and is administered by parents or teachers of children with ASD. Higher scores are indicative of greater severity. Normative data have been derived from a sample of over 1,600 children.
  A total Total-score of 76 or higher is considered severe and strongly associated with a clinical diagnosis of Autistic Disorder. T-scores of 66 through 75 are interpreted as indicating Moderate deficiencies in reciprocal social behavior that are clinically significant and lead to substantial interference in everyday social interactions, whereas T-scores of 60 to 65 are in the Mild range and indicate mild to moderate deficits in social interaction. T scores of 59 and below are considered to be within typical limits and generally not associated with clinically significant ASD.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 29 | 28
Units on a scale | -2.6 (8.3) | -6.1 (7.8)

7. Secondary Outcome: Change in Clinical Global Impression - Improvement (CGI-I) Score
Description: Measures the clinical impression of improvement on a 7-point Likert scale (ranging from 1 - very much improved - to 7 - very much worse) is a commonly used measure of overall improvement in intervention studies of children with ASD. This tool will be completed by the parent and caregiver, and is therefore considered a modified version of the instrument, which is normally completed by a clinician. This is considered an exploratory analysis of this outcome tool since it is being used in a non-standard fashion. The number of participants who "responded" in each group is the number where the parents reported that their child was improved, much improved, or very much improved.
Time Frame: Baseline, Week 6
Measure: Number; unit: # parents reporting improvement
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 29 | 28
# parents reporting improvement | 12 | 10

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: * Families advised at start of study to contact study coordinator if child experiences a new health problem.
  * Families sent weekly e-mail which includes form asking about new health problems. If "yes", study doctor contacted and reviews form and contacts participant to obtain additional info and determine if further medical evaluation/treatment required.
  AE form questions are standard questions on FDA serious adverse event (SAE) forms.
Arm/Group | Omega-3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 10/29 | 6/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 (N=29) | Placebo (N=28)
Asthma Flare (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Croup (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elective Tonsillectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrointestinal virus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased self-stimulatory behavior (Psychiatric disorders) | 1 (1) | 0 (0)
Increased tantrums (Psychiatric disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nosebleed (Vascular disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
vomitting (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No